CLINICAL TRIAL: NCT07139418
Title: Exploring the Predictive Value of Lymph Node Examination From Different Gastric Mesenteric Regions for Prognosis After D2 Lymphadenectomy Plus Complete Mesogastric Excision in Gastric Cancer Patients
Brief Title: Impact of Gastric Mesentery With Lymph Node Metastasis on Prognosis in Gastric Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: zywxm001
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Gastric Carcinoma
Keywords: Gastric cancer; Complete mesogastric excision; Gastric mesentery; Lymph node metastasis
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- D2+CME surgery for gastric cancer: D2 lymphadenectomy plus complete mesogastric excision in gastric cancer patients

SUMMARY:
This study aims to validate the predictive value of lymph node-metastasis gastric mesenteric regions and their quantitative involvement for gastric cancer prognosis by systematically examining lymph nodes from distinct mesenteric compartments in post-D2+CME radical gastrectomy specimens.

DETAILED DESCRIPTION:
Prior to 2010, the gastric cancer nodal staging systems primarily consisted of two approaches: the UICC/AJCC classification (by the International Union Against Cancer/American Joint Committee on Cancer), which was based principally on the number of metastatic lymph nodes; and the JGCA system (by the Japanese Gastric Cancer Association), which focused on the anatomical location of nodal metastases. However, a landmark unification occurred in the 14th edition of the Japanese Classification of Gastric Carcinoma (2010), where the anatomically-based nodal staging was abolished in favor of a metastasis-counting method. This harmonization with the UICC/AJCC system established a globally authoritative standard for evaluating therapeutic outcomes in gastric cancer, representing a milestone advancement in clinical research.

The current staging standard for gastric cancer follows the 8th edition TNM classification system (effective 2017) jointly established by the UICC (International Union Against Cancer) and AJCC (American Joint Committee on Cancer), which primarily evaluates tumor invasion depth (T), lymph node metastasis extent (N), and distant metastasis status (M). By integrating these three parameters, gastric cancer is classified into stages 0 through IV to guide treatment decisions and prognostic assessment. The gastric mesentery contains vascular, adipose, neural, and lymphoid tissues and can be anatomically divided into the left gastric mesentery, right gastric mesentery, left gastroepiploic mesentery, right gastroepiploic mesentery, posterior gastric mesentery, and short gastric mesentery. Although the anatomical location of metastatic lymph nodes is no longer included in the current gastric cancer staging system, our institutional research has demonstrated that among patients with the same N-stage, those with a greater number of lymph node-positive mesenteric regions exhibit worse prognosis, indicating that the anatomical distribution of nodal metastases remains clinically significant for gastric cancer outcomes. This study proposes to separately submit post-gastrectomy specimens with lymph nodes grouped by distinct mesenteric regions, with intraoperative demarcation of mesenteric boundaries during D2+CME surgery to achieve precise postoperative mesenteric sorting. Compared to the lymph node grouping method specified in the 15th edition of the Japanese Gastric Cancer Association's "Japanese Classification of Gastric Carcinoma" (2017), submitting lymph nodes according to mesenteric regions offers greater practicality. By examining gastric lymph nodes from separate mesenteric compartments, we aim to further investigate how the specific locations of lymph node-positive mesenteric regions and the total number of involved mesenteric areas impact gastric cancer patient prognosis, thereby enabling more accurate prediction of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years
2. Primary gastric adenocarcinoma confirmed by preoperative pathology result
3. cT2-4aN0-3M0 at preoperative evaluation according to the American Joint 8 Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. Patients who received gastrectomy with D2 lymphadenectomy plus complete mesogastric excision
5. American Society of Anesthesiologists (ASA) class I, II, or III
6. Written informed consent

Exclusion Criteria:

1. Negative preoperative biopsy
2. Too late tumour stage or metastasis (cT4b/M1)
3. BMI>30 kg/m2
4. Total gastrectomy or proximal gastrectomy
5. previous neoadjuvant chemotherapy or radiotherapy
6. Previous upper abdominal surgery
7. Combined with other malignant diseases
8. Reject operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the above inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | through study completion, an average of 3 year
  Prognostic impact of lymph node-positive mesenteric count in gastric cancer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xie D, Gao C, Lu A, Liu L, Yu C, Hu J, Gong J. Proximal segmentation of the dorsal mesogastrium reveals new anatomical implications for laparoscopic surgery. Sci Rep. 2015 Nov 6;5:16287. doi: 10.1038/srep16287. PMID 26542081
- [Background] Xie D, Wang Y, Shen J, Hu J, Yin P, Gong J. Detection of carcinoembryonic antigen in peritoneal fluid of patients undergoing laparoscopic distal gastrectomy with complete mesogastric excision. Br J Surg. 2018 Oct;105(11):1471-1479. doi: 10.1002/bjs.10881. Epub 2018 Jul 2. PMID 29964324
- [Background] Xie D, Liu L, Osaiweran H, Yu C, Sheng F, Gao C, Hu J, Gong J. Detection and Characterization of Metastatic Cancer Cells in the Mesogastrium of Gastric Cancer Patients. PLoS One. 2015 Nov 13;10(11):e0142970. doi: 10.1371/journal.pone.0142970. eCollection 2015. PMID 26566136
- [Background] Xie D, Shen J, Liu L, Cao B, Wang Y, Qin J, Wu J, Yan Q, Hu Y, Yang C, Cao Z, Hu J, Yin P, Gong J. Complete mesogastric excision for locally advanced gastric cancer: short-term outcomes of a randomized clinical trial. Cell Rep Med. 2021 Mar 16;2(3):100217. doi: 10.1016/j.xcrm.2021.100217. eCollection 2021 Mar 16. PMID 33763656